CLINICAL TRIAL: NCT00263952
Title: Immunotherapy of Bee Venom Allergy: Evaluation of a New Purified Bee Venom Preparation in Comparison With Already Published Studies.
Brief Title: Efficacy and Safety of a Purified Standardised Bee Venom Preparation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Al0202ig
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Bee Venom Allergy
Keywords: Bee venom allergy; Specific immunotherapy
MeSH Terms: conditions — Venom Hypersensitivity | interventions — Bee Venoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: bee venom

SUMMARY:
The trial is performed to assess efficacy and safety of a purified standardised bee venom preparation in bee venom allergy

ELIGIBILITY:
Inclusion Criteria:

* History of bee venom allergy,
* Positive RAST for bee venom,
* Positive skin prick test for bee venom

Exclusion Criteria:

* Serious chronic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-03; Primary Completion 2005-01 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Narkus, M.D., Principal Investigator
Locations (1):
- Allergopharma GmbH & Co. KG, Reinbek, Germany

REFERENCES:
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de